CLINICAL TRIAL: NCT04275245
Title: Single Center, Single Arm, Open Clinical Study to Access Safety and Initial Efficacy of Anti-CD147 Humanized Meplazumab for Injection to Treat With 2019-nCoV Pneumonia
Brief Title: Clinical Study of Anti-CD147 Humanized Meplazumab for Injection to Treat With 2019-nCoV Pneumonia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20200101
Record Dates: First submitted 2020-02-06; First posted 2020-02-19 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Coronavirus Disease 2019 (COVID-19)
Keywords: COVID-19, pneumonia
MeSH Terms: conditions — COVID-19; Pneumonia | interventions — meplazumab; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Meplazumab (Experimental): 10mg Meplazumab by intravenous infusion, every day for 2 days
  Interventions: Drug: Meplazumab for Injection

INTERVENTIONS:
Drug: Meplazumab for Injection — humanized MAb against CD147

SUMMARY:
To evaluate the safety and efficacy of humanized Meplazumab for Injection in patients infected by 2019-nCoA.

DETAILED DESCRIPTION:
According to the results of nonclinical study of humanized Meplazumab for Injection, a single dose will be used for the treatment. The treatment plan is first dose on the first day (0d) and second dose on the second day (1D) of the treatment period by intravenous(IV) infusion, each dose 10mg; The third dose will be given within 3-5 days after the second dose according to the patient's 2019-nCoV nucleic acid load, clinical manifestations and the overall evaluation of doctors, dose is 10mg. 30 mg of methylprednisolone will be given intravenously 30 minutes before each administration. Each subject will be evaluated the therapeutic effect within 28 days after the first administration, and to determine the preliminary therapeutic effect, safety and tolerability of humanized Meplazumab for Injection.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 75 years (inclusive)
* In line with the new coronavirus infection pneumonia diagnosis and treatment plan (trial version 4) issued by the Health Commission, patients with new coronavirus (2019 ncov) pneumonia were clinically diagnosed;
* The subjects must be able to understand the study and willing to participate in the study, and sign the informed consent (if the subjects with no behavioral ability think it is in their own interests to participate in the test, they should sign the informed consent by their legal guardian, or notify the consent by phone (recording) and explain it in the original medical record and other relevant documents).

Exclusion Criteria:

* Known or expected to have allergic reactions or a history of allergy to any of the ingredients treated in this trial;
* In the judgment of the investigator, there are other reasons that the patient is not suitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
2019 nCoV nucleic acid detection | 14 days
  Virological clearance rate using Real-Time PCR in upper and/or lower respiratory tract samples at day 3, day 7 and day 14 respectively.

SECONDARY OUTCOMES:
Recovery of body temperature | 14 days
  Time (days) from initiation of Meplazumab treatment until normalization of body temperature (≤37℃ axilla)
Recovery of resting respiratory rate | 14 days
  Time (days) from initiation of Meplazumab treatment until normalization of resting respiratory rate (≤24/min)
Recovery of SPO2 | 14 days
  Time (days) from initiation of Meplazumab treatment until normalization of SPO2 (>94%)
Chest CT / chest film changes | 28 days
  Rate of lung imaging recovery
PaO2 / FiO2 | 14 days
  Rate of PaO2 / FiO2 recovery
Time to reach the isolation release standard | 28 days
  Days to reach the isolation release standard
Changes of inflammatory immune status | 14 days
  Rate of CRP, D-Dimer test recovery

CONTACTS AND LOCATIONS:
Locations (1):
- Tangdu Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343